CLINICAL TRIAL: NCT03404336
Title: Pilot Randomized Controlled Trial to Evaluate the Efficacy of Well-Being Therapy Vs a Control Condition in Chronic Migraine Patients
Brief Title: Study on 30 Outpatients with Chronic Migraine Treated with Well-Being Therapy or with a Control Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Fiammetta Cosci, Associate Professor in Clinical Psychology, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBT in MIG
Record Dates: First submitted 2017-12-31; First posted 2018-01-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Chronic Migraine
Keywords: migraine; chronic; well-being therapy; psychotherapy; therapy
MeSH Terms: conditions — Migraine Disorders; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: This is a pilot study, designed as a randomized (1:1) controlled trial, comparing WBT vs a control condition. The patients will receive a baseline assessment to confirm the diagnosis of chronic migraine, then socio-demographic information, information on pharmacological/non-pharmacological treatments, on the history of medical diseases and on the psychological status will be collected as well as the number of migraine attacks per month, the duration of migraine attacks, the occurrence of migraine exclusively with menses, and the level of disability related to migraine. Thereafter, the subjects will be randomly assigned to WBT or to a control condition. The subjects will be re-assessed at the end of session 4, 8 of treatment, at 3-month and 6-month follow-ups.
Who Masked: Participant
Masking Description: Participants will not be informed if they will receive the WBT or the control condition. Of course, after the end of the study they will receive this information and they will be told why they were blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Well-being therapy (Experimental): WBT will be used as the only non-pharmacological therapeutic strategy and 8 sessions will be delivered every other week with a duration of 60 minutes each. The manualized WBT will be used (Fava, 2016). Thus, the initial phase will be concerned with self-observation of psychological well-being. Once the instances of well-being will be properly recognized, the patient will be encouraged to identify thoughts, beliefs, and behaviors leading to premature interruption of well-being (intermediate phase). The final part will involve cognitive restructuring of dysfunctional dimensions of psychological well-being and meeting the challenge that optimal experiences may entail.
  Interventions: Behavioral: Well-Being Therapy
- Control condition (Placebo Comparator): The control condition will include 8 be-weekly sessions based on Lifestyle and well-being National Institute for health and Care Excellence (NICE) guidelines (https://www.nice.org.uk/guidance/lifestyle-and-wellbeing) and on World Health Organization 12 steps to healthy eating (http://www.euro.who.int/en/health-topics/disease-prevention/nutrition/a-healthy-lifestyle). These sessions will inform participants about well-being and which lifestyles can influence it.
  Interventions: Other: Control condition

INTERVENTIONS:
Behavioral: Well-Being Therapy — Session 1: identifying and setting episodes of wellbeing into situational context. Session 2: identifying interfering thoughts and behaviors. Session 3: illustrating autonomy, reflecting and practicing it. Session 4: illustrating environmental mastery, reflecting and practicing it. Session 5: illustrating positive relations with others, reflecting and practicing it. Session 6: illustrating personal growth, reflecting and practicing it. Session 7: illustrating self-acceptance, reflecting and practicing it. Session 8: illustrating purpose in life, reflecting and practicing it.
  Arms: Well-being therapy
Other: Control condition — Session 1: illustrating the concept of lifestyle and well-being. Session 2 and session 3: illustrating healthy eating and steps to healthy eating. Session 4: illustrating physical exercise and how it promotes health. Session 5: illustrating smoking and tobacco and how they can damage health. Session 6: illustrating alcohol and how it can damage health. Session 7: illustrating drugs misuse and how it can damage health. Session 8: illustrating sexual health. No access to specific WBT ingredients will be allowed.
  Arms: Control condition

SUMMARY:
Chronic migraine is a disabling type of migraine and is often resistant to treatment. Non-pharmacological interventions have been investigated as potential treatment although, unfortunately, the literature on their efficacy is poor and showed mixed results. Well-Being Therapy (WBT) is a brief psychotherapy which has shown efficacy in decreasing the relapse rates of depression in adults, in generalized anxiety disorder and in cyclothymia. It can be implemented to empower psychological well-being. The aim of the present study is to test the efficacy of WBT in a sample of patients with chronic migraine to verify if it reduces the disability due to migraine and distress, it increases the psychological well-being as well as the level of euthymia.

DETAILED DESCRIPTION:
Chronic migraine is a disabling type of migraine and is often resistant to treatment. Non-pharmacological interventions have been investigated as potential treatment although, unfortunately, the literature on their efficacy is poor and showed mixed results. The psychological interventions tested up to now are the Acceptance and Commitment Therapy and the Mindfulness. Well-Being Therapy (WBT) is a brief psychotherapy which has been manualized in 2016 and has shown efficacy in randomized clinical trials. It showed to be effective in decreasing the relapse rates of depression in adults, it showed to be effective in generalized anxiety disorder and in cyclothymia. Thus, psychological well-being can be implemented and empowered via a specific psychotherapy and this implementation might produce a protecting effect, thus favoring prevention. The aim of the present study is to test the efficacy of WBT in a sample of patients with chronic migraine. First the efficacy of WBT will be verified in terms of disability due to migraine. Then, the efficacy of WBT will be measured in terms of psychological well-being, euthymia, and distress. For this purpose, 30 chromic migraine outpatients will be enrolled in a randomized, controlled, open clinical study.

ELIGIBILITY:
Inclusion criteria:

1. able and interested in participating to the present research project, as proved by signed Informed consent;
2. 18-65 years of age;
3. Italian mother tongue;
4. diagnosis of chronic migraine according to the International Classification of Headache Disorders. Thus, presenting specific features (i.e., unilateral and pulsating pain of moderate or severe intensity, which is aggravated or precipitated by routine physical activities and is combined with nausea and/or vomiting, photophobia, and phonophobia) and migraine headache on ≥ 15 days per month;
5. headache chronicity for a minimum of 1 year and pattern of headache symptoms stable for a period of at least 6 months;
6. no pharmacological therapy or dietary supplements use for chronic migraine OR pharmacological therapy/dietary supplement use for chronic migraine stable since at least 3 months;
7. psychotropic medication allowed only if stable since at least three months.

Exclusion criteria:

1. diagnosis of medication overuse headache;
2. co-occurrence of psychiatric disorder(s) according to the Diagnostic and Statistical Manual of mental disorders (DSM) 5th edition as diagnosed via the MINI International Neuropsychiatric Interview;
3. co-occurrence of chronic unstable medical conditions;
4. being pregnant or lactating;
5. under exogeneous hormones treatment (i.e., hormonal contraceptives, postmenopausal hormone therapy);
6. any other condition that, according to the Investigators' opinion, may alter the ability of the patient to follow study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
disability due to migraine | from baseline to 3-month follow up
  level of disability due to migraine assessed via the Migraine Disability Assessment Score (score from 0 to >21, for total score > 6 disability is clinically relevant)
frequency of migraine attacks | from baseline to 3-month follow up
  frequency of migraine attacks assessed via a daily self-report headache diary (higher the frequency, higher the severity of migraine)
duration of migraine attacks | from baseline to 3-month follow up
  duration of migraine attacks assessed via a daily self-report headache diary (higher the duration, higher the severity of migraine)
intensity of migraine attacks | from baseline to 3-month follow up
  intensity of migraine attacks assessed via a daily self-report headache diary (higher the intensity, higher the severity of migraine)

SECONDARY OUTCOMES:
level of anxiety and depression | from baseline to 3-month follow up
  the level of anxiety and depression will be assessed via the Symptom Questionnaire (total score from 0 to 92, higher is the total score and worse is the symptomatology)
level of psychological well-being | from baseline to 3-month follow up
  assessed via the World Health Organization-Five Well-Being Index (WHO 5) (total score from 0 to 25, higher total score means higher quality of life)
level of psychological well-being | from baseline to 3-month follow up
  assessed via Psychological Well-Being Questionnaire (PWB) (total score from 84 to 504, higher score corresponds to higher psychological well-being)
the level of euthymia | from baseline to 3-month follow up
  the level of euthymia will be assessed via the euthymia scale (total score from 0 to 10, higher score corresponds to higher level of euthymia)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Fiammetta COSCI, Florence, Florence
  - Centro Cefalee e Farmacologia Clinica, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mansueto G, De Cesaris F, Geppetti P, Cosci F. Protocol and methods for testing the efficacy of well-being therapy in chronic migraine patients: a randomized controlled trial. Trials. 2018 Oct 16;19(1):561. doi: 10.1186/s13063-018-2944-5. PMID 30326932